CLINICAL TRIAL: NCT01181089
Title: A Multicenter, Randomized, Blinded, Placebo-Controlled, Dose Escalation Study to Evaluate the Penetration and Pharmacodynamic Effects of Baminercept in the Cerebrospinal Fluid (CSF) and Safety in Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: Dose Escalation Study to Evaluate the Penetration and Pharmacodynamic Effects of Baminercept in the Cerebrospinal Fluid (CSF)and Safety in Subjects With Secondary Progressive Multiple Sclerosis (SPMS)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 104MS101
Record Dates: First submitted 2010-08-05; First posted 2010-08-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-01

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — baminercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Placebo
Biological: Baminercept

SUMMARY:
This is a prospective, randomized, multicenter, dose escalation study to determine subject safety, pharmacokinetic, and pharmacodynamic responses in patients with SPMS

DETAILED DESCRIPTION:
This study is a prospective, randomized, placebo-controlled, blinded, dose escalation study of 3 to 4 cohorts with defined number of patients per cohort receiving active drug or placebo for a period of 4 months followed by safety monitoring for an additional 4 months after the last dose

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Secondary Progressive Multiple Sclerosis
* Aged 18 to 57 years old, at the time of informed consent

Exclusion Criteria:

* History of clinically important (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, immune, psychiatric, hepatic, renal or hematologic insufficiency or any other major disease other than MS ( Multiple Sclerosis)
* Inability in the opinion of the Investigator to comply with study requirements
* Other protocol-defined criteria may apply

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09

PRIMARY OUTCOMES:
Measure: Change in cerebrospinal fluid levels of secondary lymphoid organs chemokines from baseline with baminercept relative to placebo | after 4 months of treatment

SECONDARY OUTCOMES:
Number of subjects experiencing Serious Adverse Event (SAE) and Adverse Event (AE) with baminercept relative to placebo | 8 months (4 months on drug, 4 months post-drug)